CLINICAL TRIAL: NCT01262794
Title: A Phase 1, Randomized, Double-blind, Placebo Controlled, Single-center, Single Dose Study to Evaluate the Safety and Tolerability, Pharmacokinetics and Pharmacodynamics of CDP6038 Administered Subcutaneously to Healthy Japanese Males
Brief Title: Pharmacokinetic (PK)/Pharmacodynamic (PD), Study of Single-dose Subcutaneous CDP6038 in Healthy Japanese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: RA0074; 2010-022543-38 (EudraCT Number)
Record Dates: First submitted 2010-12-16; First posted 2010-12-17 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteers; Japanese
MeSH Terms: interventions — olokizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- CDP6038 0.3 mg/kg (Experimental)
  Interventions: Biological: CDP6038
- CDP6038 1 mg/kg (Experimental)
  Interventions: Biological: CDP6038
- CDP6038 3 mg/kg (Experimental)
  Interventions: Biological: CDP6038
- CDP6038 6 mg/kg (Experimental)
  Interventions: Biological: CDP6038
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CDP6038 — 100 mg/mL solution for injection, single dose
  Arms: CDP6038 0.3 mg/kg; CDP6038 1 mg/kg; CDP6038 3 mg/kg; CDP6038 6 mg/kg
Biological: Placebo — 0.9% sodium chloride for injection Single-dose
  Arms: Placebo

SUMMARY:
To evaluate the safety and tolerability of CDP6038 following single dose subcutaneous (sc) administration of CDP6038 to Japanese subjects.

To evaluate the Pharmacokinetics of CDP6038 following single dose sc administration of CDP6038 to Japanese subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese volunteers

Exclusion Criteria:

* Subject has participated in any other clinical drug study (including a biologic product or a medical device) within 5 PK half-lives or 3 months (whichever is longer) prior to Screening, or the subject is currently participating in another clinical study.
* Subject is not healthy (eg, taking any drug treatments, any psychological or emotional problems, a drug/alcohol abuse or a having a history of drug/alcohol abuse, having abnormal safety parameters)

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Maximum drug concentration (Cmax) | Multiple sampling from 0 to 113 days following single dose
Area under the plasma drug concentration versus time curve from hour 0 to the time with a last quantifiable level (AUC0-t) | Multiple sampling from 0 to 113 days following single dose
Area under the plasma drug concentration versus time curve extrapolated to infinity (AUC) | Multiple sampling from 0 to 113 days following single dose
Apparent volume of distribution (Vz/F) | Multiple sampling from 0 to 113 days following single dose
Apparent total body clearance (CL/F) | Multiple sampling from 0 to 113 days following single dose
Terminal elimination half-life (T½) | Multiple sampling from 0 to 113 days following single dose

SECONDARY OUTCOMES:
PK/PD relationship between systemic CDP6038 exposure and suppression of selected acute phase markers (such as C-reactive protein), following single subcutaneous doses of CDP6038 in Japanese subjects | Multiple sampling from 0 to 15 weeks following single dose
Immunogenicity of single subcutaneous doses of CDP6038 in Japanese subjects | Multiple sampling from 0 to 15 weeks following single dose

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (1):
- Guildford, Surrey, United Kingdom